CLINICAL TRIAL: NCT02390427
Title: Phase Ib Dose-escalation Trial of Taselisib (GDC-0032) in Combination With Anti-HER2 Therapies in Participants With Advanced HER2+ Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otto Metzger, MD (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Otto Metzger, MD, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-024
Record Dates: First submitted 2015-03-11; First posted 2015-03-17 (Estimated); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Breast Cancer; Recurrent Breast Cancer
Keywords: Metastatic Breast Cancer; Advanced Breast Cancer; Recurrent Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — 2-(3-(2-(1-isopropyl-3-methyl-1H-1,2-4-triazol-5-yl)-5,6-dihydrobenzo(f)imidazo(1,2-d)(1,4)oxazepin-9-yl)-1H-pyrazol-1-yl)-2-methylpropanamide; Ado-Trastuzumab Emtansine; pertuzumab; Trastuzumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm A (Experimental): Arm A
  - Taselisib with Trastuzumab emtansine (also called T-DM1)
  * Taselisib administered orally, daily in each treatment cycle (3 weeks).
  * Trastuzumab emtansine (also called T-DM1) administered once via IV per treatment cycle (3 weeks).
  Interventions: Drug: Taselisib; Drug: Trastuzumab emtansine
- Arm B (Experimental): Arm B
  -Taselisib with T-DM1 and Pertuzumab
  * Taselisib is administered oral, daily or every other day per treatment cycle (3 weeks).
  * Trastuzumab emtansine (also called T-DM1) administered once via IV per treatment cycle (3 weeks).
  * Pertuzumab- administered once via IV per treatment cycle (3 weeks).
  Interventions: Drug: Taselisib; Drug: Trastuzumab emtansine; Drug: Pertuzumab
- Arm C (Experimental): Arm C:
  * Taselisib with Pertuzumab and Trastuzumab
  * Cohort C will not open without additional authorization from Genentech
    * Taselisib is administered oral, daily in each treatment cycle (3 weeks).
    * Trastuzumab administered once via IV per treatment cycle (3 weeks).
    * Pertuzumab- administered once via IV per treatment cycle (3 weeks).
  Interventions: Drug: Taselisib; Drug: Pertuzumab; Drug: Trastuzumab
- Arm D (Experimental): Arm D
  * Taselisib with Pertuzumab, Trastuzumab, and Paclitaxel
  * Cohort will not be opened without additional authorization from Genentech
    * Taselisib- administered oral, daily in each treatment cycle (3 weeks).
    * Pertuzumab- administered once via IV per treatment cycle (3 weeks).
    * Trastuzumab administered once via IV per treatment cycle (3 weeks).
    * Paclitaxel- administered via IV, weekly for 3 weeks within each cycle.
  Interventions: Drug: Taselisib; Drug: Pertuzumab; Drug: Trastuzumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Taselisib
  Other Names: GCD-0032
Drug: Trastuzumab emtansine
  Other Names: T-DM1; Kadcyla
  Arms: Arm A; Arm B
Drug: Pertuzumab
  Other Names: Perjeta
  Arms: Arm B; Arm C; Arm D
Drug: Trastuzumab
  Other Names: Herceptin
  Arms: Arm C; Arm D
Drug: Paclitaxel
  Other Names: Taxol; Onxal
  Arms: Arm D

SUMMARY:
This research study is a way of gaining new knowledge about the combination of Taselisib with other drugs in the treatment of metastatic breast cancer. Taselisib is an investigational drug which works by blocking a protein called PI3K (phosphoinositide 3-kinase) that helps cancer cells grow. This drug has been used in laboratory experiments and information from these studies suggests that this drug may help to prevent or slow the growth of cancer cells. The main purpose of this study is to find the appropriate dose of Taselisib to be used with other drugs in further clinical studies. This is an open-label, 3+3 dose-escalation phase Ib study to identify the Maximum Tolerated Dose(s) (MTD) and to identify the recommended phase 2 dose (RP2D) of Taselisib. This study will be conducted in 4 separate arms. (A-D).

DETAILED DESCRIPTION:
This study is divided in two parts, a combination dose finding escalation part (Part 1) and a dose combination expansion part (Part 2). Participants will enter only one Part (either 1 or 2) and receive study drugs from only one combindation of study drugs, know as arms, as assigned by the main study physician. The study includes four different arms as listed below:

* Arm A: Taselisib with Trastuzumab emtansine (also called T-DM1)
* Arm B: Taselisib with Trastuzumab emtansine and Pertuzumab
* Arm C: Taselisib with Pertuzumab and Trastuzumab
* Arm D: Taselisib with Pertuzumab, Trastuzumab, and Paclitaxel

Part 1: Since we are looking for the highest dose of Taselisib that can be administered safely without severe or unmanageable side effects in participants that have breast cancer, not everyone who participates in Part 1 of this research study will receive the same dose of the Taselisib. The dose participants get will depend on the number of participants who have been enrolled in the study before and how well they have tolerated their doses.

Each combination dose will only be given to a group of 3 - 6 participants. The results from each group will be reviewed and depending on the results, a different combination dose or schedule may be investigated in the next group of participants or the same combination dose taken by a participant may be repeated with the next group of participants to investigate these results further (a different schedule means that instead of taking doses once every day, participants may take them only on some days in the week).

Part 2: The doses in this part will be based on the best combination doses from Part 1. This part will look at the potential side effects and see how your cancer responds to the drug.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic, locally advanced , or locally recurrent breast cancer
* Histologically confirmed HER2+ invasive breast cancer
* Measurable or non-measurable disease per RECIST v1.1
* Prior therapy - Prior trastuzumab, lapatinib, pertuzumab, and trastuzumab emtansine (T-DM1) are allowed. Patients who have received prior therapy with Taselisib (GDC-0032) or BYL-719 are excluded. There is no limit on the number of prior lines of therapy.
* ECOG performance status 0 or 1
* Normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥ 1,500/mm3
  * Platelets ≥100,000/mm3
  * Total bilirubin < 1.5 X institutional upper limit of normal. For patients with Gilbert syndrome, the direct bilirubin should be within the institutional normal range
  * AST (SGOT) and ALT (SGPT) < 2.5 X institutional upper limit of normal
  * Serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 mL/min
  * Fasting glucose ≤ 120 mg/dL and HbA1c < 7%
* Left ventricular ejection fraction ≥ 50%
* Women of childbearing potential (including those who have had a tubal ligation) must have a documented negative pregnancy test within 14 days prior to planned initiation of Taselisib.
* Ability to understand and the willingness to sign a written informed consent document.
* For Part 2: patients must have tissue that is amenable to biopsy and must be willing to undergo research biopsy. Patients who undergo an attempted research biopsy procedure for the purpose of this protocol, and in whom inadequate tissue is obtained, are not required to undergo a repeat biopsy in order to continue on protocol.

Exclusion Criteria:

* Anti-cancer therapy within 2 weeks prior to entering the study or those who have not recovered from acute adverse events due to agents administered more than 2 weeks earlier. Palliative radiation to bony metastases ≥2 weeks prior to study entry is allowed.
* Prior treatment with a PI3 kinase, AKT or mTOR inhibitor in which the patient experienced a Grade ≥3 drug related adverse event or otherwise would be at increased risk for additional PI3K related toxicity
* Currently receiving any other investigational agents. Treatment with an investigational agent within 2 weeks prior to planned initiation of study therapy is allowed provided that any drug related toxicity has completely resolved
* Major surgical procedure within 4 weeks prior to planned initiation of study therapy
* Significant traumatic injury within 3 weeks prior to planned initiation of study therapy
* Known untreated brain metastases are excluded. History of treated CNS metastases is okay, provided the following criteria are met:

  * Disease outside the CNS is present.
  * No evidence of interim progression between the completion of CNS directed therapy and the screening radiographic study
  * No history of intracranial hemorrhage or spinal cord hemorrhage
  * Not requiring anti-convulsants for symptomatic control
  * Minimum of 3 weeks between completion of CNS radiotherapy and Cycle 1 Day 1 and recovery from significant (Grade ≥ 3) acute toxicity with no ongoing requirement for corticosteroid
* History of allergic reactions or hypersensitivity attributed to compounds of similar chemical or biologic composition to the Taselisib drug formulation or other agents used in this study.
* Receiving any medications or substances that are inhibitors of CYP3A4.
* Malabsorption syndrome or other condition that would interfere with enteral absorption
* Active small or large intestine inflammation such as Crohn's disease or ulcerative colitis
* Type 1 or 2 diabetes requiring anti hyperglycemic medication (e.g. metformin, glipizide, insulin)
* Leptomeningeal disease as the only manifestation of the current malignancy
* Congenital long QT syndrome or QTc > 500 msec
* Active congestive heart failure or ventricular arrhythmia requiring medication
* Uncontrolled ascites requiring weekly large volume paracentesis for 2 consecutive weeks prior to initiation of study treatment
* Active infection requiring intravenous (IV) antibiotics
* Patients requiring any daily supplemental oxygen
* Uncontrolled hypomagnesemia, hypokalemia or hypocalcemia, defined as values below the lower limit of normal (LLN) for the institution despite adequate electrolyte supplementation or management
* Symptomatic hypercalcemia requiring continued use of bisphosphonate or denosumab therapy
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* Grade ≥2 peripheral neuropathy
* Any other diseases, active or uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, pulmonary dysfunction, metabolic dysfunction, psychiatric illness/social situations, physical examination finding, or clinical laboratory finding that would limit compliance with study requirements.
* Women of childbearing potential (< 1 year amenorrheic) or sexually active males who are not employing adequate contraception (or practicing complete abstinence).

  * Female patients of childbearing potential must commit to using a reliable and appropriate method of contraception until at least 7 months after the end of last dose of study treatment.
  * Male patients with a partner of childbearing potential must agree to use a barrier method of contraception (condom) in addition to having their partner use another contraceptive method during the trial and for 7 months after the last dose of study treatment.
* Pregnant women and women who are lactating.
* Known human immunodeficiency virus (HIV) infection
* Inability or unwillingness to swallow pills

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2015-04-20 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2024-07 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Taselisib in combination with anti-HER2 therapy(ies) and/or paclitaxel. | 28 Days

SECONDARY OUTCOMES:
Clinical Benefit Rate (CBR) for efficacy of Taselisib in combination with anti-HER2 therapy(ies) and/or paclitaxel. | > or = 6 Months
  Defined as complete response (CR) + partial response (PR) + stable disease (SD) using RECIST 1.1
Progression Free Survival (PFS) for efficacy of Taselisib in combination with anti-HER2 therapy(ies) and/or paclitaxel. | 2 Years
  Defined as the time from the date of the first dose of study treatment until the date of first documentation of progressive disease (PD) or death from any cause (whichever occurs first)
Overall Survival for efficacy of Taselisib in combination with anti-HER2 therapy(ies) and/or paclitaxel. | 2 Years
  Defined as the time from the date of the first dose of study treatment until the date of death from any cause
Occurrence of AEs and SAEs during treatment with Taselisib in combination with anti-HER2 therapy(ies) and/or paclitaxel. | 2 Years
  Defined with CTCAE version 4.0
Occurrence of dose delays or holds | More than 7 Days
  Defined as a delay or hold of one of the study agents for more than 7 days
Occurrence of dose reductions | 2 Years
Dose Limiting Toxicity of Taselisib in combination with anti-HER2 therapy(ies) and/or paclitaxel. | 28 Days
  Defined as a toxicity within the DLT Assessment Window.

CONTACTS AND LOCATIONS:
Overall Officials: Otto Metzger, MD, Principal Investigator — Dana Farber Cancer Insitute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Sarah Cannon Research Institute, Nashville, Tennessee